CLINICAL TRIAL: NCT01630993
Title: Milking the Umbilical Cord at Term Cesarean Birth: Effect on Hemoglobin Levels in the First 48 Hours of Life
Brief Title: Milking the Umbilical Cord at Term Cesarean Birth
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Debra Erickson-Owens, Assistant Professor, University of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HU0708-113M
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Anemia
Keywords: umbilical cord milking; umbilical cord stripping; umbilical cord clamping; placental transfusion; placental residual blood volume
MeSH Terms: conditions — Anemia; Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Umbilical Cord Milking (Experimental): At birth, the infant will be held below the level of the placenta and umbilical cord will be milked 5 times after birth and before clamping the cord.
  Interventions: Other: Umbilical Cord Milking
- Immediate Cord Clamping (No Intervention): At birth, the infant will be held at the level of the placenta and umbilical cord will be clamped within 10 seconds (routine practice).

INTERVENTIONS:
Other: Umbilical Cord Milking — At birth, the infant will be held below the level of the placenta and umbilical cord will be milked 5 times after birth and before clamping the cord.
  Other Names: Umbilical Cord Stripping
  Arms: Umbilical Cord Milking

SUMMARY:
The purpose of this pilot study is to determine if umbilical cord milking at the time of scheduled cesarean section effects the hemoglobin and hematocrit levels of full-term infants as determined by hemoglobin and hematocrit levels at 36-48 hours of life. This study will help to establish the feasibility of umbilical cord milking as an alternative to delayed clamping at the time of planned cesarean section.

DETAILED DESCRIPTION:
New evidence suggests the practice of immediate clamping and cutting of the umbilical cord at birth may contribute to anemia in infancy. Immediate clamping can deprive a full term infant of 60 to 100 ml of whole blood representing 30 to 50 mg/kg of iron. The "low tech-low cost" intervention of delayed cord clamping can reduce anemia in infancy by enhancing placental-infant transfusion at birth. The risk of maternal bleeding makes a delay in cord clamping at the time of cesarean section challenging. In the United States (US), immediate clamping and cutting of the umbilical cord is the usual practice at the time of cesarean section. Milking of the umbilical cord may offer an alternative to delayed cord clamping for the prevention of anemia in infancy when time and speed are critical factors at the time of cesarean section. Although some obstetrical and pediatric providers fear adverse outcomes from delayed cord clamping or umbilical cord milking such as polycythemia or jaundice, the most recent clinical trials fail to support these fears.

In spite of iron supplementation and iron fortified formula and food, iron deficiency in infants and toddlers remains a significant public health problem in the US. Poor iron stores in the first year of life can lead to iron deficiency which has the potential to cause harm to the developing brain.

The number of births by cesarean section is on the rise in this country. According to the latest US birth data reported by the National Center for Health Statistics, the cesarean section rate is now above 32%, over a 50% increase since 1996. Immediate cord clamping is routine practice at the time of cesarean section in the US. Consequently over 1.4 million babies annually will have their umbilical cords cut immediately at the time of birth. This routine practice interferes in placental transfusion and results in less blood volume and red blood cells and increases anemia at birth and lowers total body iron stores in the newborn at six months. The potential effect of immediate cord clamping at cesarean section is enormous on the public health of infants in this country. However the association between cord clamping time and infant well-being is not generally recognized by clinicians.

Delaying the clamping and cutting of the cord for just two minutes is known to offer benefit and can improve the iron stores of term newborns extending into at least the first six months of life. Although there is benefit for the baby, a two minute delay is not feasible for the mother at time of cesarean section. However, milking of the umbilical cord at the time of cesarean section may be a viable alternative to delayed cord clamping and may prevent anemia and infant iron deficiency. Most of the available literature on umbilical cord milking was written over 50 years ago. Even so, these studies support the technique as safe for term infants resulting in higher neonatal hemoglobin and hematocrit levels. One recent study found cord milking was beneficial and did not cause harm in very low birth weight preterm infants.

This study will help to establish the feasibility of using umbilical cord milking as an alternative to delayed cord clamping at the time of cesarean section. Umbilical cord milking will be examined as a selective intervention to accelerate placental transfusion when delayed clamping is not ideal. It has the potential to prevent anemia and iron deficiency in infancy in full-term infants born by cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Women at full term gestation (37-41 weeks) with:
* Uncomplicated, singleton pregnancy
* English speaking
* Planning an elective Cesarean Section
* Not in labor

Exclusion Criteria:

* Major medical or obstetrical complications
* Women who smoke
* Intrauterine growth restriction
* Serious congenital anomalies

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Newborn Hemoglobin and Hematocrit levels | 36-48 hours of life
  At 36-48 hours, term infants (born by planned cesarean section) exposed to umbilical cord milking will have higher hemoglobin and hematocrit levels compared to infants exposed to immediate cord clamping

SECONDARY OUTCOMES:
Placental Residual Blood Volume | At birth
  Term infants (born by planned cesarean section) exposed to umbilical cord milking will have lower placental residual blood volume compared to infants exposed to immediate cord clamping

CONTACTS AND LOCATIONS:
Overall Officials: Debra Erickson-Owens, PhD, CNM, Principal Investigator — University of Rhode Island; Judith Mercer, PhD, CNM, Principal Investigator — University of Rhode Island and Women & Infants Hospital
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Erickson-Owens DA, Mercer JS, Oh W. Umbilical cord milking in term infants delivered by cesarean section: a randomized controlled trial. J Perinatol. 2012 Aug;32(8):580-4. doi: 10.1038/jp.2011.159. Epub 2011 Nov 17. PMID 22094494